CLINICAL TRIAL: NCT03235492
Title: Clinical Study of Salivary Glycated Albumin
Brief Title: Salivary Glycated Albumin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team did not receive the necessary study equipment from our international partners.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Chairman of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00076395
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; salivary glycated albumin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SmartAlbu (Experimental): If a participant agrees, after obtaining informed consent, the investigator will measure and record temperature, blood pressure, heart rate, height and weight. The participant will be given detailed instruction on how to hold the container and will be asked to spit (or deposit) their saliva up to the indicated line. The procedure will be performed twice to study the reproducibility of the test. The participant will then be asked to have a standard blood draw of 2-3 mls of blood into a vacutainer tube for analysis of HbA1c at the central lab and 1-2 mls of blood for glycated albumin for assay analysis, and a finger stick for point of care HbA1c measurement.
  Interventions: Device: SmartAlbu

INTERVENTIONS:
Device: SmartAlbu — Plan:
  1. Consent an individual
  2. Measure and record temperature, blood pressure, heart rate, height and weight
  3. Obtain two samples of saliva for the SmartAlbu portable salivary sensor
  4. Take a venous blood sample for HbA1c and
  5. Glycated albumin
  6. Obtain blood sample from a finger stick for point of care HbA1c device

SUMMARY:
(1) to determine whether the ratio of glycated albumin and total albumin in saliva is equivalent to blood and (2) to investigate whether the non-invasive SmartAlbu portable salivary sensor is as accurate as standard tests that measure glycosylated hemoglobin (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* 123 individuals with type 1 or type 2 diabetes
* 53 non diabetic controls
* Age: 18 to 80
* Body mass index >18.5kg / m2

Exclusion Criteria:

* Acute illness (within 7 days) - respiratory infection, fever above 38 °C, sinusitis infection, severe allergies.
* Individuals with known sickle cell, pregnancy, hemoglobinopathies, renal failure
* Subjects unable to give voluntary informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Salivary glycated albumin vs. blood glycated albumin | 30 min
  Whether the ratio of glycated albumin and total albumin in saliva is equivalent to blood.
Salivary glycated albumin vs. glycosylated hemoglobin (HbA1c) | 30 min
  To investigate whether the non-invasive SmartAlbu portable salivary sensor is as accurate as standard tests that measure HbA1c.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MBBS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No